CLINICAL TRIAL: NCT05349773
Title: The Pneumatic Tourniquet Technique for Endoscopic Radial Artery Harvest; Does it Affect Patient Hemodynamics?
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: MFM-IRB, R.22.02. 1615.R1
Record Dates: First submitted 2022-04-14; First posted 2022-04-27 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Ischemic Heart Disease; Coronary Artery Bypass Graft
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- endoscopic left radial artery harvesting: single group of 32 patients listed for coronary artery bypass surgery with endoscopic radial artery harvesting.
  Interventions: Procedure: Pneumatic tourniquet, endoscopic left radial artery harvesting

INTERVENTIONS:
Procedure: Pneumatic tourniquet, endoscopic left radial artery harvesting — Endoscopic radial artery harvesting technique is performed after applying a tourniquet over the distal arm proximally to the elbow. The tourniquet pressure is increased 90 mmHg over the systolic pressure and the tourniquet time will be monitored.
  he changes in Heart rate (HR), systolic blood pressure (SBP) and diastolic blood pressure (DBP) will be assessed before and after deflating the tourniquet every 5 minutes for 30 minutes.

SUMMARY:
This study aims to investigate the effect of the pneumatic tourniquet technique on the patients' hemodynamics; heart rate (HR), systolic blood pressure (SBP) and diastolic blood pressure (DBP).

DETAILED DESCRIPTION:
Coronary artery bypass graft surgery (CABG) is the most common cardiac surgical procedure. Radial artery of the non-dominant hand with better ulnar collaterals is preferred over the saphenous vein because of long term patency of the radial artery. Radial artery is the preferred second or third arterial conduits for vessels with sub occlusive stenosis.

There are two techniques of radial artery harvesting; open and endoscopic techniques. Endoscopic radial artery harvesting (ERAH) is increasing and it is possible but the evidence regarding its safety is scarce. ERAH is cosmetically better than the open technique.

ERAH technique is performed after applying a tourniquet over the distal arm proximally to the elbow. Allen test will be done first and if the hand has a good blood supply through the ulnar artery, the tourniquet pressure is increased 75-100 mmHg over the systolic pressure and the tourniquet time is kept under one hour and the left radial artery will be endoscopically harvested.

During the time of tourniquet inflation, there is ischemia of the forearm with subsequent cellular ischemic changes like; cellular acidosis, cellular edema, and activation of cellular apoptosis. On deflating the tourniquet, there is reperfusion of the limb and development of ischemic / reperfusion injury with a subsequent increase of inflammatory mediators and reactive oxygen species (ROS). These changes may be associated with some hemodynamic instability that might be dangerous, especially in patients with ischemic heart disease (IHD).

ELIGIBILITY:
Inclusion Criteria:

* Listed for CABG surgery with the use of ERAH technique.

Exclusion Criteria:

* Emergency CABG surgery.
* CABG plus any other cardiac surgery.
* The use of inopressor drugs before ERAH

Ages: 30 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who are listed for CABG surgery with the use of ERAH technique at cardiothoracic and vascular surgery center (Mansoura University Hospitals, Mansoura University) are eligible for this study.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
heart rate | the changes in HR are being assessed at baseline for 30 minutes and for 30 minutes of deflating the tourniquet.
  HR will be recorded at inflating the tourniquet and every five minutes for thirty minutes. HR will be recorded at tourniquet deflation and every five minutes for total of thirty minutes.
systolic blood pressure | the changes in SBP are being assessed at baseline for 30 minutes and for 30 minutes of deflating the tourniquet.
  SBP will be recorded at inflating the tourniquet and every five minutes for thirty minutes. SBP will be recorded at tourniquet deflation and every five minutes for total of thirty minutes.
diastolic blood pressure | the changes in DBP are being assessed at baseline for 30 minutes and for 30 minutes of deflating the tourniquet.
  DBP will be recorded at inflating the tourniquet and every five minutes for thirty minutes. DBP will be recorded at tourniquet deflation and every five minutes for total of thirty minutes.

SECONDARY OUTCOMES:
Phenylephrine use | The phenylephrine use ( for SBP less than 100 mmHg) will be recorded for one hour
  0 microgram of phenylephrine will be used after deflating the tourniquet if systolic blood pressure is lower than 100mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Elsayed M Abdelkarime, MD, Study Chair — Lecturer of Anesthesia and Surgical Intensive Care; Ahmed A Eisa, MD, Study Director — Lecturer of Anesthesia and Surgical Intensive Care
Locations (1):
- Mansoura University, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data will be available (including data dictionaries).
  Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will be available immediately following publication and no end date.
Access Criteria: The data will be shared with anyone who wishes to access the data. To achieve the aims in the approved proposal. Data will be available indefinitely at my research gate account under the name (Elsayed Abdelkarime)